CLINICAL TRIAL: NCT02021682
Title: CNS and Plasma Amyloid-Beta Kinetics in Alzheimers's Disease; A Blood Isotope Labeled Amyloid-beta Test for Alzheimer's Disease.
Brief Title: CNS and Plasma Amyloid-Beta Kinetics in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: In Vivo metabolism of ABeta; R01NS065667 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2013-12-27 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Alzheimer's Disease
Keywords: Aβ; ABeta; ABeta kinetics; Alzheimer's Disease; Alzheimer's; amyloid beta; biomarker; dementia; PET/PIB
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and cerebro spinal fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Amyloid positive (Amyloidosis): Amyloidosis defined by positive Positive emission tomography (PET)/Pittsburg Compound B (PIB) score, or low CSF Aβ42 concentration.
- Amyloid negative (Control): Amyloid negative defined by negative Positive emission tomography (PET)/Pittsburg Compound B (PIB) score or high/normal CSF Aβ42 concentration .

SUMMARY:
Alzheimer's disease (AD) is the most common cause of dementia and currently has no disease modifying treatments or simple accurate diagnostic tests. The goal of this project is to study how amyloid-beta (a protein thought to cause AD) is made, transported and cleared in the human body. Better understanding of these processes may lead to improved understanding of AD, earlier diagnosis and a way to evaluate treatment.

DETAILED DESCRIPTION:
The overall goal is to determine the changes that occur in amyloid-beta (Aβ) metabolism in Alzheimer's disease (AD) and model the production, transport, metabolism and clearance of Aβ in the human central nervous system (CNS) and periphery to improve clinical trial designs and also possibly develop an AD blood test.

Clearance of brain Aβ occurs by enzymatic digestion (e.g. Insulin Degrading Enzyme, Neprilysin, etc.), cellular uptake and breakdown, transport across the blood-brain-barrier, and transport from the brain to cerebrospinal fluid (CSF) and then to blood. However, the relationship between CNS Aβ and blood Aβ is not known in humans and only partly understood in other animals. The goal is to determine the kinetics of Aβ in the CNS and blood to test the hypothesis that altered Aβ kinetics in the CNS in AD is associated with altered blood Aβ labeling kinetics. Understanding blood and CSF Aβ kinetics will contribute to a better understanding of Aβ production, transport, and breakdown within and between the brain, CSF and blood compartments. These fundamental measurements of Aβ kinetics in AD will help determine the effects of peripheral Aβ metabolism on pathophysiologic changes in AD. This information will provide key insights into whole body Aβ metabolism and will be useful for understanding the causes of AD. Further, these results may lead to a specific blood biomarker for AD.

Aim 1. To determine blood Aβ isoform SILK (stable isotope-linked kinetics) using existing steady state infusion labeled blood samples from amyloid positive and amyloid negative control participants. Blood Aβ kinetics will be compared to CSF Aβ kinetics and combined utilizing multi-compartment and structural models to determine the direction and magnitude of transport and breakdown.

Current labeling methods employ a primed continuous infusion which labels Aβ to near steady-state. In order to provide additional kinetic information on Aβ kinetics and potentially better distinguish AD from controls, an alternative pulse labeling protocol is proposed. In addition to providing clearer information on Aβ transport and clearance, the simplified labeling method makes blood Aβ kinetics feasible as a clinical test for treatment trials or as a diagnostic test.

Aim 2. To perform pulse bolus labeling in amyloid positive and amyloid negative controls and measure CSF Aβ isoform kinetics and blood Aβ isoform kinetics. Participants will be recruited to complete a pulse labeling study. Results from Aim 2 will be incorporated into complimentary models with results from Aim 1 and ongoing studies to provide measures of Aβ production, transport, and breakdown within and between the brain, CSF and blood compartments.

Approach: Based on preliminary data and published studies, the hypothesis will be tested that blood Aβ isoform kinetics are disrupted in AD and to model the Aβ production, transport and clearance between the brain and periphery. The data from these studies will be useful to model the production, transport and breakdown of Aβ throughout the human body.

Results of these aims will be utilized in complimentary modeling approaches and combined with the results of prior studies to provide a comprehensive model of in vivo Aβ kinetics in both the human CNS and periphery. The data and models will be able to confirm and exclude current hypotheses of human Aβ metabolism. The goals of the aims are to determine the CNS Aβ isoform kinetics with a pulse labeling protocol (Aim 1), and to determine the peripheral blood Aβ isoform kinetics with a pulse labeling protocol (Aim 2).

Experimental Design: A pulse labeling protocol with twenty participants was completed to simplify labeling. Pulse labeling experiments provided additional kinetics results to determine Aβ kinetic models. Of the next sixty participants most will be re-enrolled that have completed prior intravenous steady-state labeling Aβ SILK studies. All participants will have had a PET/PIB scan completed for fibrillar amyloid deposition measurements or CSF Aβ42 concentration measurements.

Clinical Study: A single pulse dose of leucine will be given at the beginning of the study and blood and/or CSF will be collected for 24-36 hours.

Data Analysis: We will compare the pulse labeling blood Aβ SILK results of the amyloid positive vs. amyloid negative control group for Aβ38, Aβ40, Aβ42, and ratios of isoforms vs. tests of amyloidosis such as PET/PIB scan and/or CSF Aβ42 concentration.

ELIGIBILITY:
Inclusion Criteria:

* Member of the Memory and Aging Project at Washington University
* Clinical Dementia Rating (CDR) and PET/ PIB scores
* Age 60 or greater

Exclusion Criteria:

* Clotting disorder
* Active anticoagulation therapy
* Active infection
* Meningitis
* Recent syncope
* Currently on experimental treatment targeting Aβ or medications thought to influence Aβ production or clearance rates (benzodiazepines, muscarinic agents, or anti-epileptics)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults from the Alzheimer's Disease Research Center and Memory and Aging Project at Washington University.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Analysis of SILK blood and CSF Aβ isoforms | Sample collection 24 - 96 hours post labeling
  Analysis of SILK blood and CSF Aβ isoforms will be performed. The pulse labeling blood Aβ SILK results of the amyloid positive group will be compared with the control group for Aβ38, Aβ40, Aβ42, and ratios of isoforms vs. tests of amyloidosis such as PET/PIB scan and/or CSF Aβ42 concentration.

SECONDARY OUTCOMES:
Age | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) and Age.
CSF tau/ptau | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) for CSF tau/ptau.
PET/Fluoro-D-glucose (FDG) scan findings. | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) and by PET/Fluoro-D-glucose (FDG) scan findings.
ApoE | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) for Apolipoprotein E (ApoE).
Mutation status | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) and mutation status for AD.
Cognitive measures | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) and cognitive measures.
Clinical measures | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) and clinical measures.
MRI | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) and by Magnetic resonance imaging (MRI) findings.

OTHER OUTCOMES:
novel CSF biomarkers | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) for novel CSF biomarkers.
novel imaging protocols | Sample collection 24-96 hours post labeling
  SILK blood and CSF Aβ isoforms analyzed by clinical diagnosis (AD vs. controls) and by novel imaging protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Bateman, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD at this time

REFERENCES:
- [Background] Mawuenyega KG, Sigurdson W, Ovod V, Munsell L, Kasten T, Morris JC, Yarasheski KE, Bateman RJ. Decreased clearance of CNS beta-amyloid in Alzheimer's disease. Science. 2010 Dec 24;330(6012):1774. doi: 10.1126/science.1197623. Epub 2010 Dec 9. PMID 21148344
- [Background] Potter R, Patterson BW, Elbert DL, Ovod V, Kasten T, Sigurdson W, Mawuenyega K, Blazey T, Goate A, Chott R, Yarasheski KE, Holtzman DM, Morris JC, Benzinger TL, Bateman RJ. Increased in vivo amyloid-beta42 production, exchange, and loss in presenilin mutation carriers. Sci Transl Med. 2013 Jun 12;5(189):189ra77. doi: 10.1126/scitranslmed.3005615. PMID 23761040